CLINICAL TRIAL: NCT05564455
Title: Comparison of SRK-T With Kane Formula for Prediction of Refractive Outcome After Phacoemulsification
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUI/CTR/2022/10
Record Dates: First submitted 2022-09-29; First posted 2022-10-03 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Cataract; Surgery; Phacoemulsification; Biometry; Intraocular Lens Power
MeSH Terms: conditions — Cataract | interventions — Biometry

STUDY DESIGN:
Intervention Model Description: Prospective, interventional study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SRK-T Formula for Prediction of refraction (Active Comparator): To compare post-operative refractive outcome with Sanders Retzlaff Kraff theoretical (SRK T) and Kane formulae for intraocular lens (IOL) power calculation in cataract patients
  Interventions: Other: Biometry with SRK-T formula
- Kane Formula for Prediction of refraction (Active Comparator): To compare post-operative refractive outcome with Sanders Retzlaff Kraff theoretical (SRK T) and Kane formulae for intraocular lens (IOL) power calculation in cataract patients
  Interventions: Other: Biometry with Kane formula

INTERVENTIONS:
Other: Biometry with Kane formula — Kane formulae for intraocular lens (IOL) power calculation in cataract patients
  Arms: Kane Formula for Prediction of refraction
Other: Biometry with SRK-T formula — Sanders Retzlaff Kraff theoretical (SRK T) formulae for intraocular lens (IOL) power calculation in cataract patients
  Arms: SRK-T Formula for Prediction of refraction

SUMMARY:
Cataract is a leading cause of blindness in the world. Cataract surgery is one of the most commonly performed ocular procedures. We aim to compare the newer generation biometry formula; the Kane formula with the commonly used SRK-T formula for intraocular power calculation in uneventful phacoemulsification surgery to assess the post-operative refractive outcomes at one month post-surgery.

DETAILED DESCRIPTION:
Purpose: To compare post-operative refractive outcome with Sanders Retzlaff Kraff theoretical (SRK T) and Kane formulae for intraocular lens (IOL) power calculation in cataract patients Study Design: Prospective, interventional study Place and Duration of Study: Department of Ophthalmology, Fauji Foundation Hospital, Rawalpindi Material and Methods: A total of a 70 eyes, 35 in each group will be included in our study. The patients will be randomly divided into two groups. In cases of bilateral cataract, one eye will be included in each group for better control. IOL power calculation in Group A will be done with the SRK-T formula and in group 2 with the Kane Formula. Autokeratometry and A-scan ultrasound will be done for biometry. Inclusion criteria will be uncomplicated cataract in both genders. Exclusion criteria will be ocular trauma, uveitis, previous intraocular surgery, or any retinopathy. All patients will undergo phacoemulsification with foldable lens implantation by two experienced surgeons. Post-operative refractive outcome will be evaluated at one month after surgery. The two groups will be compared.

Results: The results will be calculated by SPSS. Conclusion: A conclusion will be drawn on the basis of our results.

ELIGIBILITY:
Inclusion Criteria:

* Senile cataract (nuclear, cortical, posterior subcapsular, mature, hypermature cataract)
* Absence of other ocular pathology causing diminished visual acuity
* patients above 40 years of age
* Astigmatism > 2.5 diopters

Exclusion Criteria:

* Retinal diseases
* Maculopathy
* Uveitis
* Complications during phacoemulsification
* Combined procedures
* Previous ocular surgery
* Trauma
* Secondary cataract

Ages: 40 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2021-06-17 (Actual); Primary Completion 2022-07-17 (Actual); Study Completion 2022-07-17 (Actual)

PRIMARY OUTCOMES:
Visual acuity (Snellen/logMAR) and refractive error (automated refraction in diopters) | 1 month post-operatively
  The visual acuity and refractive error of the patients will be measured 1 month post-operatively to compare between the two groups
Spherical equivalent in diopters | 1 hour to 1 year
  The spherical equivalent of the patients will be measured 1 month post-operatively to compare between the two groups
Post-operative refractive outcome in diopters | 1 hour to 1 year
  Post-operative refractive outcome will be compared with intended refractive outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Fauji Foundation Hospital, Rawalpindi, Punjab Province, Pakistan